CLINICAL TRIAL: NCT00607958
Title: Clinical Trial to Assess the Security of the Dose Reduction of Ritonavir in HIV-Infected Patients in Treatment With Tipranavir/Ritonavir 500/200 mg Every 12 Hours
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPVRTV_500100_IQ
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Tipranavir; ritonavir; dose reduction; inhibitory quotient
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir; Drug Tapering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): dose reduction
  Interventions: Drug: tipranavir/ritonavir (dose reduction)

INTERVENTIONS:
Drug: tipranavir/ritonavir (dose reduction) — tipranavir/ritonavir 500/100 BID

SUMMARY:
Tipranavir is a drug with a high antiretroviral activity, also in presence of major mutations in the protease gene. However, its necessity of being co-administered with 400 mg of ritonavir daily, limits its efficacy for the treatment of HIV-infected patients, due to the high incidence of gastrointestinal adverse events. Nevertheless, tipranavir plasma though concentrations were higher than the proposed minimum effective concentration for patients with previous experience with protease inhibitors (PI) in half of patients treated with tipranavir/ritonavir at 500/100 mg dose every 12 hours. Furthermore, when the number of mutations in the protease gene is limited, there are no differences in the reduction of the viral load between patients treated with tipranavir/ritonavir at 500/200 mg and 500/100 mg every 12 hours. At last, the efficacy of tipranavir treatment has been more closely related with the inhibition quotient (IQ) than with concentrations considered isolated.

Considering the previous arguments, it can be hypothesized that, basing in every subject IQ, it could be possible to identify those patients HIV-infected in treatment with tipranavir/ritonavir at 500/200 mg every 12 hours that could take advance of the reduction of ritonavir to 100 mg every 12 hours, without compromising the viral replication control. This strategy could improve the tolerability to the treatment, what could result in a better adherence and less proportion of treatment abandon due to this reason

DETAILED DESCRIPTION:
Tipranavir efficacy as a rescue treatment in HIV-infected patients was assessed in the RESIST studies, which included patients with a wide antiretroviral experience who were found in viral failure despite being on PI-based antiretroviral therapy and in which resistance test showed the presence of major mutations in the protease gene. In those studies treatment with tipranavir/ritonavir at 500/200 mg dose every 12 hours was related with a major probability of achieving undetectable viral load after a 48 weeks follow-up, compared with conventional PI (33.6% vs. 15.3%, respectively). However, tipranavir clinical efficacy can be limited by the appearance of adverse events, mainly on a gastrointestinal level, but also altering the lipid profile or elevating the transaminase plasmatic concentration.

According to the data of the BI 1182.52 study, response to tipranavir is related to its plasma trough concentration. So, concentrations higher than 20 mmol/L (10 times the IC90 adjusted by the binding to proteins of HIV PI-resistant-strains) are related with a major probability of achieving the viral replication suppression. This concentration was achieved by the 77% and the 48% of patients who received tipranavir 500 mg every 12 hours co-administered with 200 and 100 mg of ritonavir every 12 hours respectively. Furthermore, viral load diminution was similar between patients treated with 100 or with 200 mg of ritonavir every 12 hours, as long as the number of mutations was less than 20. These data states the importance of putting together virological (mutations in the protease gene) and pharmacokinetic data (trough levels) so the antiretroviral treatment benefit can be maximized. The subanalysis that included 157 patients of the BI 1182.52 study and 311 patients of the RESIST study showed that virological response in patients with treatment with tipranavir/ritonavir was better in patients with an IQ higher than 25-50.

With this data the following conclusions can be inferred: tipranavir is a drug with a high antiretroviral activity, also in presence of major mutations in the protease gene. However, its necessity of being co-administered with 400 mg of ritonavir daily, limits the efficacy for the treatment of HIV-infected patients, due to a high incidence of gastrointestinal adverse events. Nevertheless, trough levels of tipranavir was over the proposed minimum effective concentration for patients with previous experience with protease inhibitors (IP). Furthermore, as the number of mutations in the protease gene is limited, there are no differences in the reduction of the viral load between patients treated with tipranavir/ritonavir at 500/200 mg and 500/100 mg every 12 hours. At last, the efficacy of tipranavir treatment has been closely related with the inhibition quotient (IQ) than with concentrations obtained considered isolated.

Considering the previous arguments, it can be hypothesized that, basing in every subject IQ, it could be possible to identify those patients HIV-infected in treatment with tipranavir/ritonavir at 500/200 mg every 12 hours that could take advance of the reduction of ritonavir to 100 mg every 12 hours, without compromising the viral replication control. This strategy could improve the tolerability to the treatment, what could result in a better adherence and less proportion of treatment abandon due to this reason.

ELIGIBILITY:
Inclusion Criteria:

1. Age +=18 years.
2. HIV-infected patients.
3. Stable antiretroviral treatment including tipranavir/ritonavir 500/200 every 12 hours for at least 4 weeks.
4. HIV viral load <50 copies/mL for at least 12 weeks.
5. Resistance test (Genotype or Virtual Phenotype) before starting tipranavir treatment.
6. Tipranavir IQ +=60.
7. Subject able to follow the treatment period.
8. In women, negative pregnancy test or not in fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or undertaking to use a barrier contraceptive method during the study.
9. Signature of the informed consent.

Exclusion Criteria:

1. AIDS-defining illness in the last 4 weeks.
2. Suspicion of unsuitable antiretroviral treatment compliance.
3. In women, pregnancy or breastfeeding.
4. Record or suspicion of incapability to cooperate as appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with viral load <50 copies/mL | Basal, week 2, week 4, week 8, week 12 week 24, week 36 and week 48.

SECONDARY OUTCOMES:
Proportion of patients that show a tipranavir IQ >60 while treated with tipranavir/ritonavir 500/200 mg every 12 hours | Screening
Proportion of patients that maintain a tipranavir IQ >=40 while treated with tipranavir/ritonavir 500/100 mg every 12 hours | Basal, week 2, week 4, week 8, week 12 week 24, week 36 and week 48.
Change in CD4 lymphocytes count after 24 and 48 weeks' follow-up | Week 24 and week 48
Incidence and severity of adverse events after 24 and 48 weeks' follow-up | Week 24 and week 48
Change in lipid profile (total cholesterol, HDL-cholesterol. LDL-cholesterol and triglycerides) after 24 and 48 weeks' follow-up | Week 24 and week 48
Change in hepatic enzymes (AST, ALT and GGT) after 24 and 48 weeks' follow-up | Week 24 and week 48
In patients with virological failure, incidence of new mutations in the protease gene | When virological failure

CONTACTS AND LOCATIONS:
Overall Officials: Molto Jose, MD,PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain